CLINICAL TRIAL: NCT00134108
Title: Randomised Controlled Clinical Effectiveness Trial of Cognitive Behaviour Therapy (CBT) Versus Treatment as Usual (TAU) for Insomnia in Cancer Patients
Brief Title: Clinical Benefit of Cognitive Behaviour Therapy (CBT) for Insomnia in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Cancer Research UK (Other)
Organization: NHS Greater Clyde and Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C8265/A3036
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2005-10-26 (Estimated); Status verified 2003-01

CONDITIONS: Insomnia; Cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy

SUMMARY:
The purpose of this study is to conduct a formal controlled evaluation of the potential benefits of CBT for insomnia in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Meets clinical criteria for insomnia.
* Diagnosis of breast, prostate, colorectal or gynaecological cancer.
* In follow-up phase with no further anti-cancer therapy planned.

Exclusion Criteria:

* Anti-cancer chemotherapy or radiotherapy within 4 weeks of trial entry.
* Evidence of sleep apnoea or other sleep disorder.
* Evidence of untreated major depressive disorder.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Colin Espie, PhD, Principal Investigator — University of Glasgow
Locations (1):
- North Glasgow and Grampian Trusts, Glasgow and Aberdeen, United Kingdom

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811